CLINICAL TRIAL: NCT01476423
Title: Treatment of Glanzmann's Thrombasthenia: A Prospective Observational Registry
Brief Title: Observational Registry of the Treatment of Glanzmann's Thrombasthenia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3521; U1111-1122-5019 (Other: WHO)
Record Dates: First submitted 2011-10-07; First posted 2011-11-22 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Congenital Bleeding Disorder; Glanzmann's Disease
Keywords: Glanzmann's Thrombasthenia
MeSH Terms: conditions — Thrombasthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — A prospective, observational multi-national registry collecting data and evaluating the efficacy and safety of rFVIIa in patients with GT with past or present refractoriness to platelet transfusions. The registry will also collect data from a broader range of GT patients treated with systemic haemostatic treatment (with or without antifibrinolytic drugs or other agents) used in the clinics. Data collection will continue for a maximum of six years. Baseline data as well as data obtained during either bleeding episodes or invasive procedures/surgeries will be recorded in the registry.

SUMMARY:
This observational registry is conducted in Europe, Asia, Africa and the United States of America (USA).

The purpose of the registry is to evaluate the efficacy and safety of activated recombinant human factor VII (rFVIIa) during bleeding episodes and for the prevention of bleeding during invasive procedures/surgery in patients with Glanzmann's thrombasthenia (GT) with past or present refractoriness to platelet transfusions. Attention will be directed towards complications related to thrombo-embolic events and concomitant medications especially antifibrinolytics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital GT defined as patients with lifelong bleeding tendency characterised by impaired or absent platelet aggregation, impaired clot retraction and prolonged bleeding time or prolonged platelet function analyser closure time. The patient has normal platelet counts and platelet morphology. Optional diagnosis criteria are quantitative or qualitative evaluation of GP (Glycoprotein) IIb/IIIa receptor including flow cytometry and identification of gene defects
* Signed informed consent by the patient or next of kin or legally acceptable representative to collect data on treatment of a given bleeding episode or surgical event as specified in the protocol. If informed consent is provided by the next of kin or legally acceptable representative, consent must also be obtained from the patient as soon as he/she is able to do so. Informed consent must be obtained before entry of data into the registry

Exclusion Criteria:

* Patients with acquired thrombasthenic states caused by autoimmune disorders (acute or chronic) or drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with GT. There is no limit to the number of bleeding episodes or preventions of bleeding during invasive procedures/surgery that can be entered for each patient within the lifetime of the registry. Patients will receive standard care according to local practice, thus any systemic haemostatic treatment (with or without antifibrinolytic drugs or other agents) considered useful by the centres for treatment of GT, are included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2004-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
For bleeding episodes: Overall efficacy evaluated by the caregiver/patient | within 30 days of end of treatment
For surgery including invasive and dental procedures: Haemoglobin level | prior to surgery and 24 hours after surgery
For surgery including invasive and dental procedures: Overall haemostatic evaluation by the surgeon | 24 hours after surgery

SECONDARY OUTCOMES:
Changes in laboratory parameters (prothrombin time, platelet count, fibrinogen), if available | at the time of administration and two hours after the administration of rFVIIa
Adverse Events (AEs) | during treatment episodes
Serious Adverse Events (SAEs) | during treatment episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (15):
- Novo Nordisk Clinical Trial Call Center, Princeton, New Jersey, United States
- Algiers, Algeria
- Vienna, Austria
- Brussels, Belgium
- Sofia, Bulgaria
- Paris La Défense Cedex, France
- Mainz, Germany
- Budapest, Hungary
- Rome, Italy
- Alphen aan den Rijn, Netherlands
- Karachi, Pakistan
- Madrid, Spain
- Malmo, Sweden
- Zurich, Switzerland
- Crawley, United Kingdom

REFERENCES:
- [Derived] Poon MC, D'Oiron R, Baby S, Zotz RB, Di Minno G. The Glanzmann Thrombasthenia Registry: safety of platelet therapy in patients with Glanzmann thrombasthenia and changes in alloimmunization status. Haematologica. 2023 Oct 1;108(10):2855-2858. doi: 10.3324/haematol.2022.281973. No abstract available. PMID 36924249
- [Derived] Zotz RB, Poon MC, Di Minno G, D'Oiron R; Glanzmann Thrombasthenia Registry Investigators. The International Prospective Glanzmann Thrombasthenia Registry: Pediatric Treatment and Outcomes. TH Open. 2019 Sep 12;3(3):e286-e294. doi: 10.1055/s-0039-1696657. eCollection 2019 Jul. PMID 31523745
- [Derived] Di Minno G, Zotz RB, d'Oiron R, Bindslev N, Di Minno MN, Poon MC; Glanzmann Thrombasthenia Registry Investigators. The international, prospective Glanzmann Thrombasthenia Registry: treatment modalities and outcomes of non-surgical bleeding episodes in patients with Glanzmann thrombasthenia. Haematologica. 2015 Aug;100(8):1031-7. doi: 10.3324/haematol.2014.121475. Epub 2015 May 22. PMID 26001793
- [Derived] Poon MC, d'Oiron R, Zotz RB, Bindslev N, Di Minno MN, Di Minno G; Glanzmann Thrombasthenia Registry Investigators. The international, prospective Glanzmann Thrombasthenia Registry: treatment and outcomes in surgical intervention. Haematologica. 2015 Aug;100(8):1038-44. doi: 10.3324/haematol.2014.121384. Epub 2015 May 22. PMID 26001792
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com